CLINICAL TRIAL: NCT01317953
Title: Phase ⅠStudy of Oral Green Tea Extract as Maintenance Therapy for Extensive-stage Small Cell Lung Cancer
Brief Title: Oral Green Tea Extract for Small Cell Lung Cancer
Status: Available | Type: Expanded Access
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, M.D., Shandong Cancer Hospital and Institute
Other Study IDs: GTESCLC2011
Record Dates: First submitted 2011-03-17; First posted 2011-03-18 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — epigallocatechin gallate

INTERVENTIONS:
Dietary Supplement: epigallocatechin gallate — Starting dose green tea catechin extract "EGCG" 400 mg twice a day (BID) of EGCG (400 mg caps BID), second escalated dose 800 mg BID of EGCG (2x400 mg caps BID), third escalated dose 1200 mg BID of EGCG (3x400 mg),fourth escalated dose 1600 mg BID of EGCG (4x400 mg),and fifth escalated dose 2000 mg BID of EGCG (5x400 mg),
  Other Names: EGCG

SUMMARY:
The purpose of this study is to determine whether green tea extract is safe for extensive-stage small lung cancer who achieved objective tumor response after first-line therapy.

DETAILED DESCRIPTION:
Small-cell lung cancer accounts for 13 to 15% of all lung cancer and more than 60 to 70% of patients present with extensive disease (ED). Although etoposide plus cisplatin (EP) regimen has been the mainstay of ED-SCLC treatment, median overall survival is about 9 months, with 5 to 10% surviving two years and only 1% of patients achieving a long-term disease-free survival. To improve this outcome further, various attempts have been made, which included dose intensification with stem cell supports, maintenance therapy, and also searches for a better chemotherapy regimen.

Significant anticarcinogenic effects of green tea extract on various organs, such as skin, stomach, duodenum, colon, liver, pancreas, and lung in rodent models have been confirmed. Recent scientific investigations have identified the active chemical compounds in green tea designated tea polyphenols or catechins. Epigallocatechin-3-gallate (EGCG) is the major catechin in tea.An investigation about the effects of EGCG on human SCLC cells revealed that EGCG had similar anti-tumor effects on drug-sensitive (H69) and drug-resistant (H69VP) SCLC cells. Thus, the investigators conduct this phase I trial, the objectives of this trial were to study the side effects and best dose of of EGCG in treating patients with small-cell lung cancer who achieved objective tumor response after first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of small cell lung cancer
* extensive-stage disease
* Eastern Cooperative Oncology Group performance status (PS) of 0 to 2
* age18 years old
* Adequate bone marrow reserves: neutrophil (ANC) count ≥ 1500 /mm^3, platelet count ≥ 100,000 /mm^3, hemoglobin ≥ 9 g/dl
* Adequate renal function: serum creatinine ≤ 1.5 mg/dl and/or calculated creatinine clearance ≥ 60 ml/min
* Adequate hepatic function: bilirubin level ≤ 1.5 x ULN, ASAT & ALST ≤ 1.5 x ULN
* Signed written informed consent prior to study entry
* According to Response Evaluation Criteria in Solid Tumors(RECIST), patients didn't progress after first-line chemotherapy

Exclusion Criteria:

* Any condition that would hamper informed consent or ability to comply with the study protocol
* Participation in another research study in the last three months
* Known malignancy at any site other than SCLC
* Recent consumption of green tea (5 or more cups per day within one week of study enrollment)
* Pregnant and lactating women
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to EGCG

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Xindong Sun, M.D., Study Director — Shan Dong Tumor Hospital and Institute
Locations (1):
- Shan Dong cancer hospital and institute, Jinan, Shandong, China